CLINICAL TRIAL: NCT01596114
Title: Multicenter Trial Estimating the Persistence of Molecular Remission in Chronic Myeloid Leukemia After Stopping TKI
Brief Title: European Stop Tyrosine Kinase Inhibitor Study
Acronym: EURO-SKI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European LeukemiaNet (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ELN-001; 2011-000440-22 (EudraCT Number)
Record Dates: First submitted 2012-05-08; First posted 2012-05-10 (Estimated); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Chronic Myeloid Leukemia
Keywords: TKI; CML; Stopping; chronic phase; in remission
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stop treatment (Experimental): TKI treatment will be stopped in CML patients with very deep molecular responses for at least one year and at least 3 years TKI treatment
  Interventions: Other: Stopping treatment with TKI

INTERVENTIONS:
Other: Stopping treatment with TKI — stopping until loss of MMR

SUMMARY:
The EURO-SKI is a multicenter open label, uncontrolled trial estimating the persistence of molecular remission in Chronic Myeloid Leukemia (CML) patients after stopping Tyrosine Kinase Inhibitor (TKI). Main goal is the assessment of the duration of major molecular response (MMR) or better after stopping TKI therapy.

Secondary goals include:

* Identification of clinical and biological factors affecting the persistence of complete molecular remission after stopping TKI (e.g. level of Complete molecular remission (CMR), risk score, duration of TKI treatment, type of TKI pretreatment)
* Evaluation of quality of life (QoL) in patients stopping TKI
* Evaluation of medico-economic impact of stopping TKI
* Estimating the number of patients in CMR who are eligible for stopping TKI therapy by setting up a screening log
* Time to recovery of CMR There will be no randomised comparison. Based on the experience of the STIM trial (Mahon et al., Lancet Onc 2010) we expect an overall six-month molecular-relapse-free survival probability of at least 40%. An interim analysis will be performed after a pilot phase where 200 patients have been observed for at least six months. Formally, it is planned to test the null hypothesis H0: Six-month molecular relapse-free survival probability P ≤ 40% against the alternative hypothesis H1: Six-month molecular-relapse-free survival probability P > 40%. Eligible are adult CML patients in chronic phase on TKI treatment in CMR for at least one year (> 4 log reduction of BCR-ABL transcripts on IS, TKI treatment for at least 3 years, confirmed by a PCR within a standardized CMR laboratory). Clinical and biological monitoring will be performed during 3 years: Associated scientific projects are performed. Recruitment period: 2 years; follow up: 3 years. Planned patient recruitment in main phase: n=500

ELIGIBILITY:
Inclusion Criteria:

* CML in CP under treatment with TKI in first line or in second line because of toxicity to first line TKI or with TKI in combination
* Duration of TKI treatment before enrolment at least 3 years
* At least complete molecular remission MR4
* Before inclusion confirmation of CMR4 through a EUTOS-CMR laboratory
* Baseline data and documentation on treatment before study entry available
* Both sexes but fertile women only if using effective contraceptive
* Health insurance coverage
* 18 years or older

Exclusion Criteria:

* Under 18 years old
* Hospitalized patients without ability to give informed consent
* Adults under law protection or without ability to consent
* Previous or planned allogeneic stem cell transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 868 (Actual)
Dates: Start 2012-05-30 (Actual); Primary Completion 2014-12-03 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
molecular relapse-free survival | 3 years
  Evaluation of molecular relapse-free survival after stopping TKI (survival without molecular relapse defined by BCR-ABL1 > 0.1% on the IS at one time point (loss of major molecular response, MMR))

SECONDARY OUTCOMES:
Overall and progression-free survival | 3 years
  Overall and progression-free survival and the probabilities of a restart of TKI without prior molecular relapse
Treatment costs | 3 years
  Saved treatment costs / country from the time off TKI therapy considering also the more frequent PCR monitoring
QoL | 3 years
  Patient reported QoL and symptom burden over time
Time to recovery | 3 years
  Analysing the time to recovery of CMR4 after loss of MMR

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Saussele, Prof. Dr., Principal Investigator — Universitätsmedizin Mannheim, Universität Heidelberg
Locations (50):
- Czechia (6):
  - Fakultní nemocnice, Brno
  - Fakultní nemocnice Hradec Králové, Hradec Králové
  - University Hospital Olomouc, Olomouc
  - University Hospital Plzen, Pilsen
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Ústav hematologie a krevní transfuze, Prague
- Odense University Hospital, Odense, Denmark
- Helsinki University Central Hospital, Helsinki, Finland
- France (17):
  - CHU d'Angers, Angers
  - Institut Bergonié, Bordeaux
  - Université Victor Segalen, Bordeaux
  - Hôpital André Mignot, Chesnay
  - Chu Estaing, Clermont-Ferrand
  - Hôpital Claude Huriez, Lille
  - Hôpital Édouard Herriot, Lyon
  - Institut Paoli-Calmettes (IPC), Marseille
  - Centre Hospitalier Universitaire (CHU) de Nantes, Nantes
  - Hôpital de l'Archet, Nice
  - Hôpital Saint-Louis, Paris
  - Hôpital Necker-Enfants Malades, Paris
  - Hopital de la Milétrie, Centre Hospitalier Universitaire (CHU) de Poitiers, Poitiers
  - Hôpital Pontchaillou, Rennes
  - Hôpital Purpan, Toulouse
  - CHU de Tours, Tours
  - Hôpital de Brabois, Vandœuvre-lès-Nancy
- Germany (8):
  - Uniklinik RWTH, Aachen
  - Universitätsklinikum, Bonn
  - Klinikum, Chemnitz
  - Universitätsklinikum, Jena
  - Klinikum Kempten-Oberallgäu, Kempten
  - Universitätsmedizin Mannheim, Universität Heidelberg, Mannheim
  - Universitätsklinikum Giessen und Marburg GmbH, Marburg
  - MVZ Klinikum Straubing GmbH, Straubing
- University of Athens, Society of Hematology, Athens, Greece
- Netherlands (2):
  - VU Academic Medical Center, Amsterdam
  - Albert Schweitzer Hospital, Dordrecht
- Norway (4):
  - Oslo universitetssykehus HF Rikshospitalet, Oslo
  - Stavanger University Hospital, Stavanger
  - University Hospital of Northern Norway, Tromsø
  - Norwegian University of Science and Technology, Trondheim
- Instituto Português de Oncologia Francisco Gentil, Lisbon, Portugal
- Sweden (9):
  - Karoliniska Univ hospital Huddinge, Huddinge
  - Univ hospital Linköping, Linköping
  - Sunderby hospital, Luleå
  - Lunds Universitet, Lund
  - Univ hospital Örebro, Örebro
  - Karoliniska Univ sjh Solna, Stockholm
  - Länssj Sundsvall, Sundsvall
  - Norrlands Univ hospital, Umeå
  - Uppsala University hospital, Uppsala

REFERENCES:
- [Background] Richter J, Lubking A, Soderlund S, Lotfi K, Markevarn B, Sjalander A, Stenke L, Deneberg S, Ahlstrand E, Myhr-Eriksson K, Panayiotidis P, Gedde-Dahl T, Zackova D, Mayer J, Olsson-Stromberg U, Mahon FX, Saussele S, Hjorth-Hansen H, Koskenvesa P. Molecular status 36 months after TKI discontinuation in CML is highly predictive for subsequent loss of MMR-final report from AFTER-SKI. Leukemia. 2021 Aug;35(8):2416-2418. doi: 10.1038/s41375-021-01173-w. Epub 2021 Feb 15. No abstract available. PMID 33589755
- [Background] Soderlund S, Persson I, Ilander M, Guilhot J, Hjorth-Hansen H, Koskenvesa P, Richter J, Saussele S, Mustjoki S, Olsson-Stromberg U. Plasma proteomics of biomarkers for inflammation or cancer cannot predict relapse in chronic myeloid leukaemia patients stopping tyrosine kinase inhibitor therapy. Leuk Res. 2020 Mar;90:106310. doi: 10.1016/j.leukres.2020.106310. Epub 2020 Jan 23. PMID 32058176
- [Background] Bouillon AS, Ventura Ferreira MS, Awad SA, Richter J, Hochhaus A, Kunzmann V, Dengler J, Janssen J, Ossenkoppele G, Westerweel PE, Te Boekhorst PAW, Mahon FX, Hjorth-Hansen H, Isfort S, Fioretos T, Hummel S, Schemionek M, Wilop S, Koschmieder S, Saussele S, Mustjoki S, Beier F, Brummendorf TH. Telomere shortening correlates with leukemic stem cell burden at diagnosis of chronic myeloid leukemia. Blood Adv. 2018 Jul 10;2(13):1572-1579. doi: 10.1182/bloodadvances.2018017772. PMID 29980572
- [Background] Schutz C, Inselmann S, Saussele S, Dietz CT, Mu Ller MC, Eigendorff E, Brendel CA, Metzelder SK, Bru Mmendorf TH, Waller C, Dengler J, Goebeler ME, Herbst R, Freunek G, Hanzel S, Illmer T, Wang Y, Lange T, Finkernagel F, Hehlmann R, Huber M, Neubauer A, Hochhaus A, Guilhot J, Xavier Mahon F, Pfirrmann M, Burchert A. Expression of the CTLA-4 ligand CD86 on plasmacytoid dendritic cells (pDC) predicts risk of disease recurrence after treatment discontinuation in CML. Leukemia. 2017 Apr;31(4):829-836. doi: 10.1038/leu.2017.9. Epub 2017 Jan 11. PMID 28074067
- [Result] Saussele S, Richter J, Guilhot J, Gruber FX, Hjorth-Hansen H, Almeida A, Janssen JJWM, Mayer J, Koskenvesa P, Panayiotidis P, Olsson-Stromberg U, Martinez-Lopez J, Rousselot P, Vestergaard H, Ehrencrona H, Kairisto V, Machova Polakova K, Muller MC, Mustjoki S, Berger MG, Fabarius A, Hofmann WK, Hochhaus A, Pfirrmann M, Mahon FX; EURO-SKI investigators. Discontinuation of tyrosine kinase inhibitor therapy in chronic myeloid leukaemia (EURO-SKI): a prespecified interim analysis of a prospective, multicentre, non-randomised, trial. Lancet Oncol. 2018 Jun;19(6):747-757. doi: 10.1016/S1470-2045(18)30192-X. Epub 2018 May 4. PMID 29735299
- [Result] Ilander M, Olsson-Stromberg U, Schlums H, Guilhot J, Bruck O, Lahteenmaki H, Kasanen T, Koskenvesa P, Soderlund S, Hoglund M, Markevarn B, Sjalander A, Lotfi K, Dreimane A, Lubking A, Holm E, Bjoreman M, Lehmann S, Stenke L, Ohm L, Gedde-Dahl T, Majeed W, Ehrencrona H, Koskela S, Saussele S, Mahon FX, Porkka K, Hjorth-Hansen H, Bryceson YT, Richter J, Mustjoki S. Increased proportion of mature NK cells is associated with successful imatinib discontinuation in chronic myeloid leukemia. Leukemia. 2017 May;31(5):1108-1116. doi: 10.1038/leu.2016.360. Epub 2016 Nov 28. PMID 27890936
- [Result] Rinaldetti S, Pfirrmann M, Manz K, Guilhot J, Dietz C, Panagiotidis P, Spiess B, Seifarth W, Fabarius A, Muller M, Pagoni M, Dimou M, Dengler J, Waller CF, Brummendorf TH, Herbst R, Burchert A, Janbetaen C, Goebeler ME, Jost PJ, Hanzel S, Schafhausen P, Prange-Krex G, Illmer T, Janzen V, Klausmann M, Eckert R, Buschel G, Kiani A, Hofmann WK, Mahon FX, Saussele S. Effect of ABCG2, OCT1, and ABCB1 (MDR1) Gene Expression on Treatment-Free Remission in a EURO-SKI Subtrial. Clin Lymphoma Myeloma Leuk. 2018 Apr;18(4):266-271. doi: 10.1016/j.clml.2018.02.004. Epub 2018 Feb 8. PMID 29510895